CLINICAL TRIAL: NCT00407290
Title: The Impact of an Epidural Ropivacaine-Neostigmine Injection for Perineal Analgesia at the End of Labor, on Either Immediate Postpartum Perineal Pain or Development of Chronic Perineal Pain After Vaginal Delivery.
Brief Title: The Impact of an Epidural Ropivacaine-Neostigmine Injection for Perineal Analgesia at the End of Labor.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE 2005/13mai/87
Record Dates: First submitted 2006-11-14; First posted 2006-12-05 (Estimated); Last update posted 2006-12-05 (Estimated); Status verified 2006-12

CONDITIONS: Pregnancy; Vaginal Delivery
Keywords: pregnancy; vaginal delivery
MeSH Terms: interventions — Neostigmine

INTERVENTIONS:
Drug: neostigmine

SUMMARY:
Perineal pain after childbirth occurs in the majority of women (with or without episiotomy). Perineal pain can become source of chronic pain in 9%-12% of the cases. Neostigmine a cholinesterase inhibitor at a dose of 500µg combined with Sufentanil or Ropivacaine (=local anaesthetic) is an analgesic. The goal of this study is to examine the effect of the use of epidural Neostigmine for perineal analgesia at the end of the labor on acute pain and on the development of chronic pain post partum.

DETAILED DESCRIPTION:
The goal of epidural analgesia during labour is to obtain an analgesia with a minimum of "motor block". Absence of motor block at the time of the childbirth allows to decrease the rate of instrumentation (forceps, vacuum extractor). When the parturient approach complete cervical dilatation (8-10 cm), the anaesthetist must perform a last epidural injection for perineal analgesia. Generally a local anaesthetic is used (ex : Ropivacaine). Adjuvant can be associated to local anaesthetic (Sufentanil, Clonidine and more recently Neostigmine) to maximize local anaesthetic without increasing motor block.

Neostigmine, a cholinesterase inhibitor, increase concentration of acetylcholine on synaptic level and stimulate analgesic mechanisms mediated by this acetylcholine on dorsal horn of spinal cord.

Perineal pain after childbirth appears in most of the women with or without episiotomy. (Mac Arthur Am J Obst. Gynecol. 2004). This perineal pain can become source of chronic pain in 9%-12% of the cases. Neostigmine, a cholinesterase inhibitor at the dose of 500µg, combined with Sufentanil or Ropivacaine (=local anaesthetic) has an analgesic effect.

The goal of this study is to examine the effect of epidural Neostigmine for perineal analgesia at the end of the labour and on the development of chronic pain post-partum.

Inclusion criteria : any parturient of 18-45 years, normal pregnancy, at full term and having an effective epidural anaesthesia during labour.

Exclusion criteria : multiple pregnancy, obstetric pathology, refusal of participation.

Randomisation : 2 groups of 30 patients

Method :

Installation of the epidural catheter :

- Injection of Ropivacaïne + Sufentanil

Perineal analgesia :

* Ropi Group : epidural injection of Ropivacaine
* Neostigmine Group : epidural injection of Ropivacaine and Neostigmine

Evaluation of VAS, vital signs of parturient and fetal heart rate, instrumentation rate.

Evaluation of immediate post-partum pain (48hours) and use of analgesic medication in the ward.

Evaluation of chronic pain after 10 days and 1 month.

ELIGIBILITY:
Inclusion Criteria:

* any parturient of 18-45 years
* normal pregnancy
* at full term
* having an effective epidural anesthesia during labor

Exclusion Criteria:

* multiple pregnancy
* obstetric pathology
* refusal of participation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2006-03; Study Completion 2006-10

PRIMARY OUTCOMES:
acute pain (VAS)
chronic pain (questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Roelants, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Brusssels, Belgium